CLINICAL TRIAL: NCT06902220
Title: Effectiveness of Oscillation on Postoperative Pulmonary Complications After Elective Postcardiac Surgery: a Study Protocol for a Multicenter Randomized Controlled Trial
Brief Title: Effectiveness of Oscillation on Postoperative Pulmonary Complications After Elective Postcardiac Surgery
Status: Not yet recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Southeast University, China (Other)
Responsible Party: Principal Investigator, Jingyuan,Xu, professor, Southeast University, China
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: 2024ZDSYLL381-Y01
Record Dates: First submitted 2025-03-24; First posted 2025-03-30 (Actual); Last update posted 2025-03-30 (Actual); Status verified 2024-10

CONDITIONS: Postoperative Pulmonary Atelectasis
Keywords: postcardiac surgery; oscillation; postoperative pulmonary complications
MeSH Terms: conditions — Pulmonary Atelectasis

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- Intervention group (Experimental): Once patients' CPOT score reaches 0, intubated patients will receive continuous high-frequency oscillation (CHFO) therapy three times daily, with 8-hour intervals and 10-minute sessions. Extubated patients will receive CHFO and continuous positive expiratory pressure (CPEP) therapy twice daily, with 12-hour intervals and 10-minute sessions.
  Interventions: Device: continuous high-frequency oscillation therapy
- Control group (No Intervention): Participants in the control group will only receive standard medical, nursing, and allied healthcare, with daily decisions made without the use of protocols. This includes spontaneous breathing and awakening trials as decided by the attending intensivist, ad hoc management of pain and delirium, and once or twice daily passive and active exercises determined by the physiotherapist, with patients typically remaining in bed if on ventilation.

INTERVENTIONS:
Device: continuous high-frequency oscillation therapy — Once patients' CPOT score reaches 0, intubated patients will receive continuous high-frequency oscillation (CHFO) therapy three times daily, with 8-hour intervals and 10-minute sessions. Extubated patients will receive CHFO and continuous positive expiratory pressure (CPEP) therapy twice daily, with 12-hour intervals and 10-minute sessions.
  Arms: Intervention group

SUMMARY:
Our study aims to evaluate the effectiveness of continuous high-frequency oscillation therapy in reducing PPCs in patients following elective cardiac surgery. Through a prospective, multicenter, randomized controlled trial, we seek to establish evidence that could lead to improved postoperative pulmonary care and outcomes for cardiac surgery patients.

ELIGIBILITY:
Inclusion Criteria:

* Adult patients (18 years or older) undergoing elective cardiac surgery will be included. Participants must provide informed consent upon ICU admission and have at least one risk factor for PPCs, including age ≥ 75 years, American Society of Anesthesiologists (ASA) score ≥ 2, history of chronic obstructive pulmonary disease (COPD) stage ≥ 2 or asthma (moderate to severe), current heavy smoking or heavy smoking history within the past 6 months, obstructive sleep apnea, frailty index > 0.21 or body max index (BMI) ≥ 30 kg/m².

Exclusion Criteria:

* Patients will be excluded if they have contraindications for oscillation treatment (e.g., untreated tension pneumothorax); have pneumothorax or air leak syndrome at entry; require more than 2 μg/kg/min of norepinephrine; have been diagnosed with pneumonia within 2 weeks prior to surgery; have refractory arrhythmia at entry; have a left ventricular ejection fraction < 35%; have mean pulmonary artery pressure (mPAP) > 35 mmHg; are postoperative from spinal surgery within the past 2 weeks; require a ventricular assist device; have renal failure requiring continuous renal replacement therapy (CRRT) at entry; are planned for re-operation within 48 hours or have undergone organ transplantation.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Gender Based: Yes — 18 years or older
Enrollment: 470 (Estimated)
Dates: Start 2025-09-01 (Estimated); Primary Completion 2027-01-01 (Estimated); Study Completion 2027-01-31 (Estimated)

PRIMARY OUTCOMES:
The primary outcome is the pulmonary complication severity score within 7 postoperative days, or hospital discharge, whichever came sooner. | within 7 postoperative days
  The severity of PPCs within 7 postoperative days will be assessed using an ordinal scale from 0 to 5, based on a modified definition of PPCs. Grade 0 indicated no symptoms, grade 4 represented reintubation or invasive mechanical ventilation for 48 hours or more and grade 5 indicated death before hospital discharge. PPCs occurrence and severity will be evaluated daily until 7 postoperative days or hospital discharge, using the worst score during the hospital stay for the primary analysis. Bedside chest radiographs will be performed on the first postoperative day, followed by echocardiograms on the second and third days, in addition to those requested by attending physicians.

SECONDARY OUTCOMES:
incidence of > 48 hours invasive mechanical ventilation | within 7 postoperative days
duration of mechanical ventilation | within 7 postoperative days